CLINICAL TRIAL: NCT02791880
Title: Genomic and Biomarker Predictors of Acute Kidney Injury and Other Post-Procedural Outcomes Following Transcatheter Aortic Valve Replacement
Brief Title: Acute Kidney Injury Genomics and Biomarkers in TAVR Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Amanda A Fox, MD, MPH, Professor of Anesthesiology, University of Texas Southwestern Medical Center
Other Study IDs: STU 112015-015
Record Dates: First submitted 2016-02-19; First posted 2016-06-07 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Chronic; Heart Failure; Myocardial Infarction; Arrhythmias, Cardiac; Stroke
Keywords: acute kidney injury; transcatheter aortic valve replacement; genomics; biomarker
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Heart Failure; Myocardial Infarction; Arrhythmias, Cardiac; Stroke | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA collected before procedure. Paired urine, serum, and plasma samples collected before valve replacement, six hours after valve replacement, and post-procedure days 1 and 2. Additional samples are collected on post-procedure days 3, 4 and 5 if the patient develops acute kidney injury after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TAVR patients: The group of interest is the patient population with aortic stenosis who are undergoing transcatheter aortic valve replacement (TAVR)
  Interventions: Procedure: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement — The investigators will collect blood and urine samples from patients with aortic stenosis who are undergoing transcatheter aortic valve replacement.

SUMMARY:
In the last decade, transcatheter aortic valve replacement (TAVR) has become an increasingly utilized alternative procedure for replacing a stenotic aortic valve. This study collects clinical information, DNA, blood and urine samples (throughout procedural hospitalization) in order to investigate the incidence of acute kidney injury (AKI) in patients undergoing TAVR and to identify key clinical and procedural predictors of AKI. This study seeks to identify blood and urine biomarkers that can be used for early detection of AKI around the time of the procedure. The study seeks to assess for novel genetic variants associated with development of AKI after TAVR. Finally the study seeks to assess for novel genetic variants and biomarkers that are associated with adverse cardiovascular events after TAVR and to further explore how these events may inter-relate with acute kidney injury.

DETAILED DESCRIPTION:
This study enrolls patients who have aortic stenosis who undergo TAVR at the University of Texas Southwestern Medical Center University Hospital. Development of post-TAVR AKI defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) SCr based criteria will be ascertained. Patients will be followed during primary hospitalization and during the 5 years following TAVR for adverse kidney outcomes as well as potentially related adverse cardiovascular outcomes. Clinical and procedural data is collected for each study patient. All subjects will have paired blood and urine collection done pre-TAVR, 6 hours after aortic valve prosthesis deployment, and on post-procedure days 1 and 2. Subjects who develop AKI will also have paired blood and urine samples collected on days 3, 4 and 5. Patients receive follow-up questionnaires by mail or email asking about hospitalizations as well as visits to cardiology, nephrology and primary care physicians. Questionnaires will also ask about health-related quality of life using validated study questionnaires. Patient follow-up will occur at regular intervals until 5 years after TAVR procedure.

ELIGIBILITY:
Inclusion criteria: Subjects are eligible to participate if they are undergoing TAVR for aortic stenosis at the University of Texas Southwestern Medical Center.

Exclusion Criteria:

1. The patient cannot or will not provide informed consent.
2. The patient is aged less than 18 years.
3. The patient's pre-procedural hematocrit is less than 25%.
4. The patient has known human immunodeficiency virus infection
5. The patient has known hepatitis C that has not been treated with antiviral medications
6. In the opinion of the principal investigator, the patient will be unlikely to complete long-term follow up for medical or social reasons (this includes transient patients and patients who have no fixed address).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from the population of patients with aortic stenosis undergoing TAVR. Enrollment will likely occur over a 15 year time period to reach target enrollment. A total of 3,000 subjects are presently targeted for enrollment at University of Texas Southwestern University Hospitals and Parkland Health and Hospital Systems.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury using KDIGO criteria | Day of procedure to post procedure day 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include serum creatinine

SECONDARY OUTCOMES:
Chronic renal insufficiency (i.e. number of patients that will have received a diagnosis of chronic renal insufficiency) | Day of procedure to year 5
  Chronic renal insufficiency is defined as patient having impaired renal function (albumin/creatinine ratio >/= 300 mg/g and eGFR <60 mL/min/1.73^2).
Heart failure per NYHA class II, III, IV | Day of procedure to year 5
  This will be measured in accordance to New York Heart Association Guidelines.
Presence of Arrhythmia (i.e. number of patients who develop an arrhythmia from postoperative day 0 to 5 years). | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post-procedural EKG reports and progress notes.
Myocardial Infarction (i.e. number of participants who develop a MI during postoperative day 0 to year 5) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post-procedural EKG reports, cardiac enzyme values, progress notes, and cardiac catheterization reports.
Cerebrovascular accident (i.e. number of participants who develop transient ischemic attack or permanent stroke during postoperative day 0 up to 5 years) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post procedural imaging data and progress notes.
Vascular complications (i.e. number of participants who develop arterial injury, dissection, limb ischemia during postoperative day 0 up to year 5) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include post procedural imaging data, progress notes and operative reports.
Need for dialysis (e.g. number of participants who undergo post-procedural dialysis) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include progress notes, and consultation notes.
Mortality (i.e. number of participants who are deceased during postoperative day 0 up to year 5) | Day of procedure to year 5
  Data will be collected from electronic medical records; data points to be collected for this measurement include progress notes and death notes.
KCCQ Quality of Life Survey | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  The Kansas City Cardiomyopathy Questionnaire (KCCQ Short Form) is a health-related quality of life measure for heart failure.
SAQ Quality of Life Survey | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  The Seattle Angina Questionnaire (SAQ Short Form) is a health-related quality of life measure for coronary artery disease.
SF12 Quality of Life Survey | Administered once prior to the procedure and 1 month to 5 years after hospital discharge
  12-item short form Health survey (SF12) is a health-related quality of life measure of functional health and well-being from the patient's point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda A Fox, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - Parkland Health & Hospital Systems, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - William J. Clements University Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
There is a possibility that individual participant data and samples will be de-identified and shared with other cohort study investigators for purposes of replicating biomarker and genetic associations with adverse outcomes.
Supporting Information: SAP, CSR
Time Frame: Data will become available at the discretion of the sponsor/Dr. Fox. Once enough data has been gathered and analyzed, and the need or DUA requests from other cohort researchers is received.
Access Criteria: Data will be collected in REDCap, a data management tool used primarily for research and QI. It is a secure, HIPAA-compliant web application. Content is backed up offsite nightly and hosted in a secure environment maintained by UTSW Information Resources. Other cohort researchers will access survey questionnaires via the secure and confidential REDCap webpage with specific view only access. Patient confidentiality is of paramount importance. Data sent outside of UTSW will be de-identified or coded. The "key" to the code (i.e. patient identifying information) will not be provided to the recipient unless a limited dataset is approved for sharing via a data use agreement between Dr. Fox/UTSW and the recipient scientist/recipient scientist's institution.

REFERENCES:
- [Background] Stortecky S, Brinks H, Wenaweser P, Huber C, Pilgrim T, Windecker S, Carrel T, Kadner A. Transcatheter aortic valve implantation or surgical aortic valve replacement as redo procedure after prior coronary artery bypass grafting. Ann Thorac Surg. 2011 Oct;92(4):1324-30; discussion 1230-1. doi: 10.1016/j.athoracsur.2011.05.106. Epub 2011 Aug 31. PMID 21880298
- [Background] Elhmidi Y, Bleiziffer S, Deutsch MA, Krane M, Mazzitelli D, Lange R, Piazza N. Acute kidney injury after transcatheter aortic valve implantation: incidence, predictors and impact on mortality. Arch Cardiovasc Dis. 2014 Feb;107(2):133-9. doi: 10.1016/j.acvd.2014.01.002. Epub 2014 Feb 17. PMID 24556191
- [Background] Giordana F, D'Ascenzo F, Nijhoff F, Moretti C, D'Amico M, Biondi Zoccai G, Sinning JM, Nickenig G, Van Mieghem NM, Chieffo A, Dumonteil N, Tchetche D, Barbash IM, Waksman R, D'Onofrio A, Lefevre T, Pilgrim T, Amabile N, Codner P, Kornowski R, Yong ZY, Baan J, Colombo A, Latib A, Salizzoni S, Omede P, Conrotto F, La Torre M, Marra S, Rinaldi M, Gaita F. Meta-analysis of predictors of all-cause mortality after transcatheter aortic valve implantation. Am J Cardiol. 2014 Nov 1;114(9):1447-55. doi: 10.1016/j.amjcard.2014.07.081. Epub 2014 Aug 13. PMID 25217456
- [Background] Thongprayoon C, Cheungpasitporn W, Srivali N, Ungprasert P, Kittanamongkolchai W, Greason KL, Kashani KB. Acute kidney injury after transcatheter aortic valve replacement: a systematic review and meta-analysis. Am J Nephrol. 2015;41(4-5):372-82. doi: 10.1159/000431337. Epub 2015 Jun 19. PMID 26113391
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Najjar M, Salna M, George I. Acute kidney injury after aortic valve replacement: incidence, risk factors and outcomes. Expert Rev Cardiovasc Ther. 2015 Mar;13(3):301-16. doi: 10.1586/14779072.2015.1002467. Epub 2015 Jan 16. PMID 25592763
- [Background] Tomey MI, Gidwani UK, Sharma SK. Cardiac critical care after transcatheter aortic valve replacement. Cardiol Clin. 2013 Nov;31(4):607-18, ix. doi: 10.1016/j.ccl.2013.07.006. PMID 24188224
- [Background] Bagur R, Webb JG, Nietlispach F, Dumont E, De Larochelliere R, Doyle D, Masson JB, Gutierrez MJ, Clavel MA, Bertrand OF, Pibarot P, Rodes-Cabau J. Acute kidney injury following transcatheter aortic valve implantation: predictive factors, prognostic value, and comparison with surgical aortic valve replacement. Eur Heart J. 2010 Apr;31(7):865-74. doi: 10.1093/eurheartj/ehp552. Epub 2009 Dec 27. PMID 20037180
- [Background] Konigstein M, Ben-Assa E, Banai S, Shacham Y, Ziv-Baran T, Abramowitz Y, Steinvil A, Leshem Rubinow E, Havakuk O, Halkin A, Keren G, Finkelstein A, Arbel Y. Periprocedural bleeding, acute kidney injury, and long-term mortality after transcatheter aortic valve implantation. Can J Cardiol. 2015 Jan;31(1):56-62. doi: 10.1016/j.cjca.2014.11.006. Epub 2014 Nov 11. PMID 25547551
- [Background] Goldberg R, Dennen P. Long-term outcomes of acute kidney injury. Adv Chronic Kidney Dis. 2008 Jul;15(3):297-307. doi: 10.1053/j.ackd.2008.04.009. PMID 18565480
- [Background] Haase-Fielitz A, Haase M, Bellomo R, Dragun D. Genetic polymorphisms in sepsis- and cardiopulmonary bypass-associated acute kidney injury. Contrib Nephrol. 2007;156:75-91. doi: 10.1159/000102072. PMID 17464117
- [Background] Bolstad BM, Irizarry RA, Astrand M, Speed TP. A comparison of normalization methods for high density oligonucleotide array data based on variance and bias. Bioinformatics. 2003 Jan 22;19(2):185-93. doi: 10.1093/bioinformatics/19.2.185. PMID 12538238
- [Background] Khawaja MZ, Williams R, Hung J, Arri S, Asrress KN, Bolter K, Wilson K, Young CP, Bapat V, Hancock J, Thomas M, Redwood S. Impact of preprocedural mitral regurgitation upon mortality after transcatheter aortic valve implantation (TAVI) for severe aortic stenosis. Heart. 2014 Nov;100(22):1799-803. doi: 10.1136/heartjnl-2014-305775. Epub 2014 Aug 25. PMID 25155800
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Movafagh S, Raj D, Sanaei-Ardekani M, Bhatia D, Vo K, Mahmoudieh M, Rahman R, Kim EH, Harralson AF. Hypoxia Inducible Factor 1: A Urinary Biomarker of Kidney Disease. Clin Transl Sci. 2017 May;10(3):201-207. doi: 10.1111/cts.12445. Epub 2017 Feb 9. PMID 28181420